CLINICAL TRIAL: NCT04794790
Title: Pilot Study to Look at Feasibility of Testing and Treatment of Combination Fentanyl and Opioid Dependent Individuals With Different Buprenorphine Induction Methods
Brief Title: Buprenorphine Induction for Fentanyl Dependent Opioid Users
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to enroll--patients uninterested in trying buprenorphine.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Kawasaki, Assistant Professor, Department of Psychiatry and Behavioral Health, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016153
Record Dates: First submitted 2021-03-01; First posted 2021-03-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Opioid Dependence Fentanyl
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: We are attempting to characterize the particular problem of prolonged precipitated withdrawal in individuals with fentanyl dependence through a quasi-experimental study, which will enroll 20 to 30 individuals at the PPI OTP, who are using fentanyl and/or combination of fentanyl and opioids but desiring buprenorphine naloxone induction. There will be a standard treatment arm, then a micro dose and macro dose arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Dose (No Intervention): Standard dose induction Visit 1 Day 1 (intake/baseline) Participants will commence induction with a dose of 4mg if COWS is above 7. If COWS is below 7, participant will be instructed to return the next day, so that COWS can be above 7 to start the study.
- Macro or High Dose (Experimental): Macro or High Dosing Visit 1 Day 1 (intake/baseline) Participants will commence induction with a dose of 4mg if COWS is above 7. If COWS is below 7, participant will be instructed to return the next day, so that COWS can be above 7 to start the study. (These participants can still be in the study and will only have to re-do a baseline COW's on the day they come back to the clinic, which will then be considered their day 1).
  Interventions: Drug: Buprenorphine/naloxone
- Micro or Low Dose (Experimental): Micro or Low Dose Visit 1 Day 1 (intake/baseline) Participants will commence induction with a dose of 4mg if COWS is above 7. If COWS is below 7, participant will be instructed to return the next day, so that COWS can be above 7 to start the study. (These participants can still be in the study and will only have to re-do a baseline COW's on the day they come back to the clinic, which will then be considered their day 1).
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Buprenorphine/Naloxone induction via a standard dose protocol
  Arms: Macro or High Dose; Micro or Low Dose

SUMMARY:
The overall goal of this pilot study is to characterize illicit fentanyl and combination fentanyl and opioid dependence explicitly, by assessing physiologic barriers to effective buprenorphine induction. Results from this pilot study may make a case for a larger feasibility study to be conducted through the Clinical Trials Network at the National Institutes of Drug Abuse.

The primary hypothesis is that individuals dependent on illicit fentanyl and combination fentanyl and opioids will have difficulty with standard buprenorphine induction, and will need a modified approach. The primary outcome measure will be retention on buprenorphine at seven days post induction. The secondary outcome measures will be objective precipitated withdrawal and the rate of patients requiring or requesting to initiate methadone due to intolerance of buprenorphine.

DETAILED DESCRIPTION:
Illicit synthetic fentanyl is found in increasing proportions of illicit drug samples, and negatively influences how buprenorphine is used on the street to help with subjective withdrawal symptoms. In the clinic, it has been observed among individuals positive for fentanyl that initiation of buprenorphine is difficult. When spontaneous withdrawal, normally the signal that the patient is ready to initiate buprenorphine, and buprenorphine is given, withdrawal symptoms often seem to increase. It is unclear whether this represents precipitated withdrawal versus progressing spontaneous withdrawal, but the standard clinical approach has been to wait for more withdrawal symptoms and time to elapse before trying another test dose. In this population, waiting is a clinically problematic strategy as many patients in continuing withdrawal would resume opioid use rather than try buprenorphine again. To date, there has been one study noting that fentanyl dependent patients are retained at equal rates to patients with heroin dependence, but this study was observational, retrospective and small. An alternative approach to induction would rapidly provide high doses of buprenorphine initially. The theory behind rapid induction would be either that the robust withdrawal observed is actually spontaneous withdrawal, calling for a higher initial buprenorphine dosing regimen, or that some of the withdrawal observed may be precipitated, but rapidly and fully occupying the receptors with partial agonist produces enough agonist effect to subdue precipitated withdrawal. If found to be superior to standard induction, the high dose induction regimen could be immediately implemented in primary care settings. Or, if buprenorphine cannot be initiated for a given patient, a full opioid agonist, namely methadone, may be the best first step, suggesting methadone as a first-line treatment for those dependent on fentanyl and other high potency synthetics. Methadone administration is currently restricted to specially licensed opioid treatment programs and not widely available across clinical settings where buprenorphine can be initiated. If the availability of methadone rescue in this study proves useful, it would support a larger case for regulatory reforms to make methadone more widely available beyond traditional OTPs.

The study proposed here would be the first pilot study to assess the extent that synthetic opioid dependence prevents successful induction with buprenorphine-naloxone. Programs like the Pennsylvania Psychiatric Institute's opioid treatment program have been set up to serve rural and impoverished small urban communities that have become the epicenter of the opioid epidemic. The need to deliver evidence-based treatment effectively is paramount, especially during a window of time in which an individual desiring treatment and having access to that treatment is vanishingly small. A difficult initiation with substantial withdrawal symptoms can derail motivation that can lead to treatment abandonment. A rapid assessment of whether individuals cannot complete buprenorphine-naloxone induction who have been using illicit fentanyl or combination fentanyl with other opioids is a starting point to change management of this growing set of individuals.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of opioid use disorder (OUD) as determined through routine clinical care
3. Positive for fentanyl on point of care urine drug screen
4. Ability to read, write, and comprehend English
5. Patients willing to start buprenorphine at the onset of treatment (e.g., clinical intake)
6. Patients who need to initiate a buprenorphine induction at home must have an operating smartphone or tablet device with video capability.

Exclusion Criteria:

1. Initiating maintenance treatment that does not include MAT or switching to a maintenance treatment that does not include MAT (i.e.: detoxification and counseling treatment only without MAT, or planning to enter methadone treatment).
2. Judged by the evaluating physician or allied clinician to need a higher level of care (i.e.: residential or inpatient treatment)
3. Pregnant
4. Patients desiring to start methadone or naltrexone at the onset of treatment (e.g., clinical intake)
5. Patients who are unable to stay in the clinic for the induction period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Number of patients on Buprenorphine at the end of 7 day induction period | 7 days
  Number of patients who are able and willing to receive a prescription for Buprenorphine at the end of a 7 day induction period. This will be measured by manual counts. The patient will be scored as 0 (for not able/willing to receive a prescription for bup) or 1 (for able/willing to receive a prescription for bup)

SECONDARY OUTCOMES:
Opioid withdrawal assessment | 7 days
  Opioid withdrawal assessment as measured by COW's and SOW's. The COWS assessment is on a 0-48 point scale, with scores of 5 or higher indicating mild or greater withdrawal symptoms. SOWS is on a 0-30 point scale, with scores of greater than 1 indicating mild withdrawal symptoms.

OTHER OUTCOMES:
Attrition rate measures | 7 days
  A measure of attrition rate. This will be assessed through manual counts either by the patient verbally stating their intention to withdraw from the study or wishing to initiate Methadone treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania Psychiatric Institute, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mars SG, Rosenblum D, Ciccarone D. Fentanyl: the many challenges ahead. Addiction. 2019 May;114(5):785-786. doi: 10.1111/add.14587. Epub 2019 Mar 15. No abstract available. PMID 30873700
- [Background] Silverstein SM, Daniulaityte R, Martins SS, Miller SC, Carlson RG. "Everything is not right anymore": Buprenorphine experiences in an era of illicit fentanyl. Int J Drug Policy. 2019 Dec;74:76-83. doi: 10.1016/j.drugpo.2019.09.003. Epub 2019 Sep 25. PMID 31563098
- [Background] Hser YI, Saxon AJ, Huang D, Hasson A, Thomas C, Hillhouse M, Jacobs P, Teruya C, McLaughlin P, Wiest K, Cohen A, Ling W. Treatment retention among patients randomized to buprenorphine/naloxone compared to methadone in a multi-site trial. Addiction. 2014 Jan;109(1):79-87. doi: 10.1111/add.12333. Epub 2013 Oct 9. PMID 23961726